CLINICAL TRIAL: NCT00084929
Title: The National CT Colonography Trial: Multicenter Assessment of Accuracy for Detection of Large Adenomas and Cancers in a Healthy Screening Population
Brief Title: The National CT Colonography Trial
Acronym: ACRIN6664
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000367101; ACRIN-6664 (Other: CIP); U01CA079778 (NIH); U01CA080098 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: colon cancer; rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT Colonography (Experimental): CT colonography conducted during the same assessment as colonoscopy.
  Interventions: Procedure: CT Colonography

INTERVENTIONS:
Procedure: CT Colonography — CT colonography performed for comparison with colonoscopy results performed during the same screening assessment.
  Other Names: CT colonography trial; colonoscopy

SUMMARY:
RATIONALE: New diagnostic procedures such as computed tomographic colonography may improve the ability to detect colorectal cancer and may provide a less invasive method of detection.

PURPOSE: This clinical trial is studying how well computed tomographic colonography works in screening healthy participants for colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the sensitivity of computed tomographic colonography (CTC) vs colonoscopy for detecting significantly large lesions (≥ 10 mm in diameter) in asymptomatic participants, in terms of specificity, area under the ROC curve, and predictive values for detecting clinically significant colorectal neoplasia.

Secondary

* Determine the interobserver variation in accuracy of interpreting CTC examinations of these participants, including any benefits of a primary 3-dimensional read and/or independent second interpretations.
* Determine the effects of different colon preparations on the accuracy of CTC in these participants.
* Compare participant acceptance and willingness to have a repeat examination by CTC vs colonoscopy.
* Determine the accuracy of CTC in detecting flat lesions in the colon of these participants.

OUTLINE: This is a multicenter study.

Participants receive an oral laxative, oral bisacodyl, and three doses of oral barium sulphate 24 hours before imaging. After cathartic cleansing, participants undergo computed tomographic colonography followed by colonoscopy.

Participants are followed up for approximately 4 weeks.

PROJECTED ACCRUAL: A total of 2,607 participants will be accrued for this study.

ELIGIBILITY:
1. Inclusion Criteria

   * Male or female outpatients
   * Aged 50 years or older
   * Scheduled for screening colonoscopy
   * Participant's signed informed consent
2. Exclusion Criteria

   * Symptoms of disease of the lower gastrointestinal tract, including

     * Melanotic stools or/and hematochezia on more than one occasion in the previous six months
     * Lower abdominal pain that would normally require a medical evaluation
   * Inflammatory bowel disease and/or familial polyposis syndrome
   * Serious medical conditions that would increase the risk associated with colonoscopy or are so severe that screening would have no benefit
   * Pregnancy
   * Previous colonoscopy within the past five years
   * Anemia (hemoglobin less than 10 gm/dl)
   * Positive fecal occult blood test (FOBT)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2600 (Actual)
Dates: Start 2005-02; Primary Completion 2007-09-11 (Actual); Study Completion 2010-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Daniel Johnson, MD, Study Chair — Mayo Clinic
Locations (14):
- United States (14):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - Invision/Radiology Imaging Associates - Englewood, Englewood, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Clinical Radiologists, S.C. at Memorial Medical Center, Springfield, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Mallinckrodt Institute of Radiology at Washington University Medical Center, St Louis, Missouri
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Researchers may request data from the ACRIN data access committee by reviewing the information at:
  https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- [Background] Vanness DJ, Knudsen AB, Lansdorp-Vogelaar I, Rutter CM, Gareen IF, Herman BA, Kuntz KM, Zauber AG, van Ballegooijen M, Feuer EJ, Chen MH, Johnson CD. Comparative economic evaluation of data from the ACRIN National CT Colonography Trial with three cancer intervention and surveillance modeling network microsimulations. Radiology. 2011 Nov;261(2):487-98. doi: 10.1148/radiol.11102411. Epub 2011 Aug 3. PMID 21813740
- [Result] Johnson CD, Herman BA, Chen MH, Toledano AY, Heiken JP, Dachman AH, Kuo MD, Menias CO, Siewert B, Cheema JI, Obregon R, Fidler JL, Zimmerman P, Horton KM, Coakley KJ, Iyer RB, Hara AK, Halvorsen RA Jr, Casola G, Yee J, Blevins M, Burgart LJ, Limburg PJ, Gatsonis CA. The National CT Colonography Trial: assessment of accuracy in participants 65 years of age and older. Radiology. 2012 May;263(2):401-8. doi: 10.1148/radiol.12102177. Epub 2012 Feb 23. PMID 22361006
- [Result] Hara AK, Blevins M, Chen MH, Dachman AH, Kuo MD, Menias CO, Siewert B, Cheema JI, Obregon RG, Fidler JL, Zimmerman P, Horton KM, Coakley KJ, Iyer RB, Halvorsen RA Jr, Casola G, Yee J, Herman BA, Johnson CD. ACRIN CT colonography trial: does reader's preference for primary two-dimensional versus primary three-dimensional interpretation affect performance? Radiology. 2011 May;259(2):435-41. doi: 10.1148/radiol.11100250. Epub 2011 Mar 1. PMID 21364081
- [Result] Hara AK, Kuo MD, Blevins M, Chen MH, Yee J, Dachman A, Menias CO, Siewert B, Cheema JI, Obregon RG, Fidler JL, Zimmerman P, Horton KM, Coakley K, Iyer RB, Halvorsen RA Jr, Casola G, Johnson CD. National CT colonography trial (ACRIN 6664): comparison of three full-laxative bowel preparations in more than 2500 average-risk patients. AJR Am J Roentgenol. 2011 May;196(5):1076-82. doi: 10.2214/AJR.10.4334. PMID 21512073
- [Result] Siewert B, Gareen I, Vanness D, et al.: ACRIN 6664: patient acceptance and preferance of CT colonography compared to optical colonoscopy for colon cancer screening. [Abstract] J Clin Oncol 27 (Suppl 15): A-4034, 2009.
- [Result] Johnson CD, Chen MH, Toledano AY, Heiken JP, Dachman A, Kuo MD, Menias CO, Siewert B, Cheema JI, Obregon RG, Fidler JL, Zimmerman P, Horton KM, Coakley K, Iyer RB, Hara AK, Halvorsen RA Jr, Casola G, Yee J, Herman BA, Burgart LJ, Limburg PJ. Accuracy of CT colonography for detection of large adenomas and cancers. N Engl J Med. 2008 Sep 18;359(12):1207-17. doi: 10.1056/NEJMoa0800996. PMID 18799557
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/types/colorectal/research/virtual-colonoscopy-results-qa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2600 asymptomatic, out-patients, 50 years or older and prescheduled for screening colonoscopy were recruited for CTC between February 2005 and December 2006.
Pre-assignment Details: Of the 2607 registration events, 7 were registration errors [duplicate registrations due to system errors] and were cancelled. Therefore, a total of 2600 unique participants were enrolled to the study.
Period: Overall Study
Arm/Group | CT Colonography
Started | 2600
Completed | 2531
Not Completed | 69
Not completed — ineligible - medical contraindication | 1
Not completed — ineligible - Pre-scheduled procedure not | 1
Not completed — Ineligible - Medical history | 6
Not completed — Withdrawal by Subject | 10
Not completed — Missing/incomplete CTC exam | 9
Not completed — Missing Reference Standard (Colonoscopy) | 42

BASELINE CHARACTERISTICS:
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1326
  Male | 1205
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97
  Not Hispanic or Latino | 2430
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10
  Asian | 54
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 325
  White | 2075
  More than one race | 20
  Unknown or Not Reported | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Advanced Adenomas (>=10mm) as Determined by Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=10mm (as measured at pathology) RS-: No Advanced adenomas >=10mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Groups:
- CT Colonography: CT colonography conducted during the same assessment as colonoscopy. CT Colonography: CT colonography performed for comparison with colonoscopy results performed during the same screening assessment.
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+ | 109
  RS- | 2422
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis Receiver-operating-characteristic (ROC) curves were estimated with the use of data pooled from the radiologists because of the small number of positive cases reviewed by each radiologist; Test type: Other; Area Under the Curve (AUC) = 0.89, 95% CI 2-sided [0.853 to 0.933]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity, for each radiologist, was calculated as the percentage of patients with lesions that were larger than or equal to the prespecified threshold and that were detected on both colonoscopy and CT colonography. The per-patient sensitivity, specificity, positive predictive value, and negative predictive value were first estimated for each radiologist, and then the average values among the radiologists were calculated; Test type: Other; Sensitivity: P(T+|D+) = 0.9, 95% CI 2-sided [0.838 to 0.96] — Exact 95% confidence intervals were calculated for each radiologist, and large-sample 95% confidence intervals were calculated for overall estimates, with the use of standard errors that allowed for estimation of variation among radiologists
Statistical Analysis 3: Comparison: CT Colonography; Specificity, for each radiologist, was calculated as the percentage of patients who did not have lesions larger than the prespecified threshold on colonoscopy as well as CT colonography The per-patient sensitivity, specificity, positive predictive value, and negative predictive value were first estimated for each radiologist, and then the average values among the radiologists were calculated; Test type: Other; P(T-|D-) = 0.86, 95% CI 2-sided [0.813 to 0.9] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV) the positive predictive value was calculated as the percentage of patients with CT colonographic findings that were also seen on colonoscopy; Test type: Other; P(D+|T+) = 0.23, 95% CI 2-sided [0.194 to 0.273] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV) the negative predictive value was calculated as the percentage of patients with no CT colonographic findings larger than the prespecified threshold that were not detected on colonoscopy; Test type: Other; P(D-|T-) = 0.99, 95% CI 2-sided [0.990 to 0.998] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants With Advanced Adenomas (>=9mm) Detected by CT Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=9mm (as measured at pathology) RS-: No Advanced adenomas >=9mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+: Advanced Adenoma >=9mm | 120
  RS-: Not Advanced Adenoma >=9mm | 2411
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"; Test type: Other; Area Under the Curve (AUC) = 0.89, 95% CI 2-sided [0.853 to 0.93]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"; Test type: Other; Sensitivity: P(T+|D+) = 0.9, 95% CI 2-sided [0.832 to 0.96] — Sensitivity indicates the percent of patients who had a lesions (of the specified size) detected by optical colonoscopy, which were detected by CTC
Statistical Analysis 3: Comparison: CT Colonography; Specificity CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"; Test type: Other; P(T-|D-) = 0.86, 95% CI 2-sided [0.817 to 0.902] — Specificity indicates the percent of patients who had not lesions detected on optical colonoscopy, who had no lesions detected on CTC
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV) CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"; Test type: Other; P(D+|T+) = 0.25, 95% CI 2-sided [0.209 to 0.292]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV) CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"; Test type: Other; P(D-|T-) = 0.99, 95% CI 2-sided [0.990 to 0.998]

3. Primary Outcome: Number of Participants With Advanced Adenomas (>=8mm) Detected by CT Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=8mm (as measured at pathology) RS-: No Advanced adenomas >=8mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+: Advanced Adenoma >=8mm | 154
  RS-: Not Advanced Adenoma >=8mm | 2377
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis; Test type: Other; Area Under the Curve (AUC) = 0.88, 95% CI 2-sided [0.842 to 0.913]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity; Test type: Other; Sensitivity: P(T+|D+) = 0.87, 95% CI 2-sided [0.803 to 0.929] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: CT Colonography; Specificity; Test type: Other; P(T-|D-) = 0.87, 95% CI 2-sided [0.825 to 0.909] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV); Test type: Other; P(D+|T+) = 0.31, 95% CI 2-sided [0.256 to 0.355]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV); Test type: Other; P(D-|T-) = 0.99, 95% CI 2-sided [0.984 to 0.994]

4. Primary Outcome: Number of Participants With Advanced Adenomas (>=7mm) Detected by CT Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=7mm (as measured at pathology) RS-: No Advanced adenomas >=7mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+: Advanced Adenoma >=7mm | 174
  RS-: Not Advanced Adenoma >=7mm | 2357
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis; Test type: Other; Area Under the Curve (AUC) = 0.87, 95% CI 2-sided [0.833 to 0.902]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity; Test type: Other; Sensitivity: P(T+|D+) = 0.84, 95% CI 2-sided [0.776 to 0.912] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: CT Colonography; Specificity; Test type: Other; P(T-|D-) = 0.87, 95% CI 2-sided [0.831 to 0.914] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV); Test type: Other; P(D+|T+) = 0.35, 95% CI 2-sided [0.299 to 0.397]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV); Test type: Other; P(D-|T-) = 0.99, 95% CI 2-sided [0.980 to 0.992]

5. Primary Outcome: Number of Participants With Advanced Adenomas (>=6mm) Detected by CT Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=6mm (as measured at pathology) RS-: No Advanced adenomas >=16mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+: Advanced Adenoma >=6mm | 210
  RS-: Not Advanced Adenoma >=6mm | 2321
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis; Test type: Other; Area Under the Curve (AUC) = 0.84, 95% CI 2-sided [0.810 to 0.878]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity; Test type: Other; Sensitivity: P(T+|D+) = 0.78, 95% CI 2-sided [0.711 to 0.849] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: CT Colonography; Specificity; Test type: Other; P(T-|D-) = 0.88, 95% CI 2-sided [0.840 to 0.92] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV); Test type: Other; P(D+|T+) = 0.4, 95% CI 2-sided [0.335 to 0.463]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV); Test type: Other; P(D-|T-) = 0.98, 95% CI 2-sided [0.971 to 0.984]

6. Primary Outcome: Number of Participants With Advanced Adenomas (>=5mm) Detected by CT Colonoscopy (Per Patient)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard (RS) for determining the existence of advanced adenomas.
  RS+: Colonoscopy found at least 1 Advanced adenomas >=5mm (as measured at pathology) RS-: No Advanced adenomas >=5mm found by colonoscopy (as measured at pathology)
Time Frame: within 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | CT Colonography
Number analyzed (Participants) | 2531
Participants
  RS+: Advanced Adenoma >=5mm | 282
  RS-: Not Advanced Adenoma >=5mm | 2249
Statistical Analysis 1: Comparison: CT Colonography; Accuracy: ROC analysis; Test type: Other; Area Under the Curve (AUC) = 0.8, 95% CI 2-sided [0.763 to 0.828]
Statistical Analysis 2: Comparison: CT Colonography; Sensitivity; Test type: Other; Sensitivity: P(T+|D+) = 0.65, 95% CI 2-sided [0.579 to 0.727] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: CT Colonography; Specificity; Test type: Other; P(T-|D-) = 0.89, 95% CI 2-sided [0.851 to 0.923] — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: CT Colonography; Positive Predictive Value (PPV); Test type: Other; P(D+|T+) = 0.45, 95% CI 2-sided [0.389 to 0.513]
Statistical Analysis 5: Comparison: CT Colonography; Negative Predictive Value (NPV); Test type: Other; P(D-|T-) = 0.95, 95% CI 2-sided [0.941 to 0.965]

7. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=10mm) Detected by CT Colonoscopy (Per Lesion)
Description: Pathology results from Colonoscopy performed up to 30 days after a CTC examination were used as the reference standard for determining the existence of advanced adenomas. CTC lesions needed to be within 2 segments and 50% size of the lesions removed via colonoscopy to be considered "detected"
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Groups:
- CT Colonography (Per Lesion): CT colonography conducted during the same assessment as colonoscopy. CT Colonography: CT colonography performed for comparison with colonoscopy results performed during the same screening assessment.
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 128
lesions
  Detected by CTC | 108
  Not Detected | 20
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion (>=10mm)); Test type: Other; Sensitivity: P(T+|D+) = 0.84, Standard Error of Mean 0.043 — Sensitivity indicates the percent of lesions in patients who had a lesions (of the specified size) detected by optical colonoscopy, which were detected by CTC

8. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=9mm) Detected by CT Colonoscopy (Per Lesion)
Description: as for outcome 7
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 143
lesions
  Detected by CTC | 117
  Not Detected | 26
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion (>=9mm)); Test type: Other; Sensitivity: P(T+|D+) = 0.82, Standard Error of Mean 0.042 — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=8mm) Detected by CT Colonoscopy (Per Lesion)
Description: as for outcome 7
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 187
lesions
  Detected by CTC | 149
  Not Detected | 38
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion >=8mm); Test type: Other; Sensitivity: P(T+|D+) = 0.8, Standard Error of Mean 0.041 — [estimate comment as in outcome 7, analysis 1]

10. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=7mm) Detected by CT Colonoscopy (Per Lesion)
Description: as for outcome 7
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 220
lesions
  Detected by CTC | 165
  Not Detected | 55
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion >=7mm); Test type: Other; Sensitivity: P(T+|D+) = 0.75, Standard Error of Mean 0.042 — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=6mm) Detected by CT Colonoscopy (Per Lesion)
Description: as for outcome 7
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 270
lesions
  Detected by CTC | 189
  Not Detected | 81
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion >=6mm); Test type: Other; Sensitivity: P(T+|D+) = 0.7, Standard Error of Mean 0.046 — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: Number of Advanced Adenoma or Cancer Lesions (>=5mm) Detected by CT Colonoscopy (Per Lesion)
Description: as for outcome 7
Time Frame: within 30 days
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | CT Colonography (Per Lesion)
Number analyzed (Participants) | 2531
Number analyzed (lesions) | 374
lesions
  Detected by CTC | 221
  Not Detected | 153
Statistical Analysis 1: Comparison: CT Colonography (Per Lesion); Sensitivity (per lesion >=5mm); Test type: Other; Sensitivity: P(T+|D+) = 0.59, Standard Error of Mean 0.045 — [estimate comment as in outcome 7, analysis 1]

13. Secondary Outcome: Interobserver Sensitivity Variability
Description: Evaluate interobserver variability in Sensitivity (P(T+|D+)) and 95% CI) when interpreting CTC examinations Each study was randomly assigned to be read independently using either a primary 2D search method (conventional 2D image display with 3D endoluminal problem solving), or a primary 3D search method (including the capability of displaying multiplanar 2D) and without prior knowledge of the colonoscopy results. A second trained radiologist of similar skill was assigned to read the images using the other modality Readers were then classified as high performing or not high performing
Time Frame: at baseline
Population: 15 readers read the 2531 case and their sensitivity was calculated as well as the variability (95% CI) in Sensitivity within 2 reader groups: High performing (HP) and not high performing (NHP). HP readers had both a sensitivity and specificity of > 85% for detecting polyps 10 mm and larger, NHP did not.
Measure: Mean (95% Confidence Interval); unit: probability of (test+ given disease+)
Units Other Than Participants: Readers
Groups:
- High Performance (HP) Readers: Readers were divided into two groups: HP readers had both a sensitivity and specificity of > 85% for detecting polyps 10 mm and larger while NHP readers had a sensitivity and/or specificity < 85%.
- Non-high Performance (NHP) Readers: NHP readers had a sensitivity and/or specificity < 85%.
Arm/Group | High Performance (HP) Readers | Non-high Performance (NHP) Readers
Number analyzed (Participants) | 2531 | 2531
Number analyzed (Readers) | 8 | 7
probability of (test+ given disease+) | 0.94 [0.825 to 0.987] | 0.88 [0.864 to 0.901]

ADVERSE EVENTS:
Time Frame: The adverse event reporting period for this protocol is defined as the period from the initiation of the Computed Tomography Colonography (CTC) procedure and self-reported events were collected for 30 days after the last primary intervention. All participants were monitored for 30days.
Description: Grade 3 Expected and Unexpected AEs with attribution of possible, probable, or definite - Routine Grade 4 Expected AEs with attribution of possible, probable, or definite - Routine Grade 4 Unexpected AEs with attribution of possible, probable, or definite Expedited Report.
  Grade 5 AEs, or Deaths with attribution of possible, probable, or definite Telephone Report and Expedited Report
Groups:
- Colonoscopy: Colonoscopy conducted during the same assessment as CT colonography
Arm/Group | CT Colonography | Colonoscopy
All-Cause Mortality (participants affected / at risk) | 0/2600 | 0/2600
Serious Adverse Events (participants affected / at risk) | 0/2600 | 1/2600
Other Adverse Events (participants affected / at risk) | 0/2600 | 0/2600
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT Colonography (N=2600) | Colonoscopy (N=2600)
hemorrhage with surgery (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalization for observation of post-polypectomy bleeding. No transfusion required.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No